CLINICAL TRIAL: NCT04841005
Title: Investigation of the Effect of Square-Step Exercise Applied by Telerehabilitation on Cognitive Functions, Balance and Quality of Life in COPD Patients
Brief Title: Investigation of Square Step Exercise Applied by Telerehabilitation in Chronic Obstructive Pulmonary Disease Patients
Acronym: COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Alp Ozel, MSc,Research assistant, Abant Izzet Baysal University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AIBU-FTR-AO-01
Record Dates: First submitted 2021-04-02; First posted 2021-04-12 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-02

CONDITIONS: COPD; Cognitive Impairment; Balance; Distorted
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Exercises will be applied with the telerehabilitation method to the individuals included in the study. Video and audio communication will be provided by free and widely used programs such as Whatsapp or Telegram. Pulse oximetry, tripod and exercise material will be given to each individual included in the study by the researcher. Individuals included in the study will be randomly divided into two groups. Exercises in both groups will be done 3 days a week for 8 weeks. Before and after each exercise session, the heart rate and oxygen saturation values of the patients will be measured by pulse oximetry, and their perception of dyspnea and leg fatigue according to the Borg scale will be recorded. The first and last evaluation of individuals will be done face to face.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Square-Step Exercise group (Experimental): Square-step exercise for 8 weeks will be applied under the supervision of a physiotherapist.
  Interventions: Other: The Square-Step Exercise Training
- Strengthening Exercise Group (Experimental): Strengthening exercise for 8 weeks will be applied under the supervision of a physiotherapist.
  Interventions: Other: Strengthening Exercise Training

INTERVENTIONS:
Other: The Square-Step Exercise Training — The Square-Step Exercise is instructed to walk according to the step pattern shown on a 100 * 250 cm mat, divided into 40 squares of 25 cm each. It includes forward, backward, lateral and diagonal steps, and step patterns are progressively made more complex. Each pattern consists of two to 16 steps; Individuals are asked to repeat the step pattern until they reach the end of the mat. Each step pattern is repeated 4-10 times to ensure that individuals can complete the pattern. The individuals included in the study will exercise in easy-difficulty patterns for the first 2 weeks, medium-difficulty patterns in the 3rd and 4th weeks, medium and advanced patterns in the 5th and 6th weeks, and advanced patterns in the 7th and 8th weeks. The square-step exercise group will perform 15 minutes of warm-up exercise, 30 minutes of progressive square-step exercise, and 10 minutes of cool-down exercise accompanied by a physiotherapist, 3 days a week.
  Arms: Square-Step Exercise group
Other: Strengthening Exercise Training — Thera-Band brand elastic bands will be used to apply resistance in strengthening training. To determine the intensity of the exercise, the perceived difficulty level after 15 repetitions with the elastic band will be evaluated with the Borg scale. If the perceived difficulty level is at the level of 12-14 (slightly difficult), it will be considered as the starting difficulty level.In the strengthening exercise group will perform, shoulder abduction, shoulder press after elbow flexion, horizontal abduction, punching with an elastic band, triceps strengthening, external rotation of the shoulder, hip abduction with external rotation and sit-to-stand exercises for 8 weeks, 3 days / week , 3 sets / sessions, 8-12 repetitions. For each exercise, it will be applied as 8 repetitions in the initial workload. In the next exercise sessions, the number of repetitions will be increased until the patient can comfortably perform 12 repetitions with the same load.
  Arms: Strengthening Exercise Group

SUMMARY:
COPD is a progressive disease associated with systemic inflammation, with many extrapulmonary outcomes such as cognitive impairment. Most of the daily activities involve doing several tasks at the same time, such as walking while talking or avoiding obstacles.

DETAILED DESCRIPTION:
The most prominent independent risk factor for cognitive impairment in COPD patients is reduced oxygen availability as a result of lung dysfunction. The prevalence of cognitive impairment in COPD patients ranges from 10% to 61%. A wide variety of tools have been developed for screening cognitive functions. The most widely used tests covering multiple cognitive domains are the Mini Mental State Examination (MMSE) and the Montreal Cognitive Assessment (MoCA).

When two tasks are performed at the same time, they compete for sources of attention, resulting in decreased performance on one or two tasks. Balance or postural control is a complex skill required for independent mobility and preventing falls. Balance performance naturally decreases with age; however, certain conditions are associated with more pronounced and rapid declines. Balance problems and fall risk are increased in COPD patients.From this perspective aim of this study is to assess the effect of square-step exercise and strengthening exercise applied with telerehabilitation on cognitive status and balance in patients with COPD.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with mild / moderate COPD by Bolu Abant Izzet Baysal University Faculty of Medicine, Department of Chest Diseases.
* Mini mental score is 23 or higher
* Being between the ages of 50-80
* Spirometric evaluation result is forced expiratory volume at one second / Forced vital capacity <70% and airflow restriction is 50% forced expiratory volume at one second <80% (expected) degree compared to post-bronchodilator forced expiratory volume at one second.
* No drug change or antibiotic use due to acute exacerbation for at least three weeks

Exclusion Criteria:

* Individuals who need continuous oxygen support
* Individuals with partial pressure of carbon dioxide≥70 mmHg
* Having a history of uncontrolled illness that may affect cognitive skills
* Have uncorrected vision and hearing impairment
* Having kyphoscoliosis and/or severe postural impairment
* Having additional risk factors (stroke, neurological disease, dementia, depression, postural hypotension, diaphragm dysfunction)

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2021-04-06 (Actual); Primary Completion 2022-02-15 (Actual); Study Completion 2022-02-15 (Actual)

PRIMARY OUTCOMES:
Change of the point in the cognitive test | Two measurements: At the beginning and after eight weeks
  Montreal Cognitive Assessment will be used to evaluate cognitive impairment. The application time of the single-page scale is approximately 10 minutes and includes 6 cognitive functions.Cognitive functions evaluated in the scale are as follows: 1. Memory 2. Visual-spatial skills 3. Executive functions, 4. Attention, concentration and working memory tasks, 5. Language, 6. Orientation. The lowest score that can be obtained from the scale is 0, the highest score is 30.
Measurement of change in postural stability | Two measurements: At the beginning and after eight weeks
  Postural stability is assessed using the Biodex Balance System. It consists of a mobile platform with 20 degrees of inclination in all directions and 12 levels of difficulty. With this system, balance is evaluated thanks to circular platforms that can oscillate simultaneously in the general, front-rear and left-right axes. The right-left stability indices are derived from the platform angular displacement in the frontal plane, while the anteroposterior angular displacement represents the platform displacement in the sagittal plane.
Measurement of change in functional balance | Two measurements: At the beginning and after eight weeks
  The Balance Evaluation Systems Test (BESTest) will be used to evaluate functional balance. BESTest examines the balance in 6 sections in order to reveal whether the special balance control systems, which are defined as biomechanical structures, stability limits / verticality, intuitive postural adjustments, postural responses, sensory orientation and walking stability, function adequately. Since some of the tasks of BESTest have two subtitles, right side and left side, the patient is evaluated under 36 titles in total. In a sequential scale where each title is scored at 4 levels, 0 represents the worst performance, 3: the best performance. The total score of the test, which has a maximum of 108 points, can be calculated separately by calculating the percentage at the end of each section, as well as calculating the percentage of the total score.
Measuring change in quality of life | Two measurements: At the beginning and after eight weeks
  St George's Respiratory Questionnaire (SGRQ) has been the most widely used quality of life measurement designed to evaluate the quality of life in lung diseases. SGRQ has distinctive (able to distinguish between different severity levels between patients) and descriptive (can detect disease progression and changes with treatment). The score range ranges from 0 (excellent health) to 100 (most severe disease) and the minimum clinically significant change is considered to be 4 units. This survey has good reproducibility in the short term. It consists of 50 questions in total. The numerical evaluation of the questionnaire is calculated in 4 separate sections as symptom score, activity score, impact score and total score.
Hospital Anxiety and Depression Scale | At the enrollment process
  It was developed to screen mood disorders in groups with a medical illness. It is a scale filled by the patient. It consists of 14 items. Substances contain 4 properties. Depression and anxiety are tried to be evaluated with the help of two subscales. The 7-item depression subscale has a scoring system between 0 and 21. The threshold value indicates "Normal" between 0-7, "Mild" between 8-10, "Moderate" between 11-14, "Severe" between 15-21.

SECONDARY OUTCOMES:
Assessment of the COPD | At the enrollment process
  COPD Assessment Test (CAT) consists of 8 questions. It was developed to reveal how patients' quality of life is affected by COPD. Each question is scored from 0 to 5, with a total score between 0 and 40. Score 0 represents the best 40 points the worst health condition. The questions were intended to cover the patients' shortness of breath, cough, sputum spitting and wheezing, as well as systemic symptoms such as fatigue and sleepiness.
Assessment of comorbidities | At the enrollment process
  The Charlson Comorbidity Index is a widely used index in many disease groups in which many potential comorbidity variables are evaluated and the relative risk is measured by giving different scores. The index consists of 19 different items. These scores given to comorbid diseases are determined according to the relative risk values of the diseases.
Evaluation of shortness of breath | At the enrollment process
  The Modified Medical Research Council Dyspnoea Scale contains 5 statements about patients' dyspnea and categorizes their dyspnea level into a 0-4 point category. Evaluates shortness of breath and activity limitation in patients
1 Minute Sit and Stand Test | Two measurements: At the beginning and after eight weeks
  The ability to stand up from a chair is an important component of maintaining independence among seniors, as this movement depends on stability and balance. The 1-minute get up and sit test is performed with a 46 cm high chair as standard, without an armrest. After the start command, it is checked whether a sit-to-sit sequence is obtained to stand up and sit from each chair. The number of cycles performed exactly after 1 minute makes up the score.
Forced expiratory volume in the first second | At the enrollment process
  Forced expiratory volume in the first second (FEV1)
Forced vital capacity | At the enrollment process
  Forced vital capacity (FVC)
The ratio of FEV1 to FVC | At the enrollment process
  The ratio of FEV1 to FVC
Mini mental test | At the enrollment process
  Although this test has limited specificity in terms of differentiating clinical syndromes, it is a short, useful and standardized method that can be used to determine the cognitive level globally. It consists of eleven items grouped under five main headings: orientation, attention and calculation, memory, and language. The test is evaluated over a total score of 30. The total score is obtained by summing the points the patient obtains from each item. The cut-off score for mild and moderate dementia in our country is calculated as 23.

CONTACTS AND LOCATIONS:
Overall Officials: Alp Özel, MSc, Principal Investigator — BAIBU, Faculty of Health Sciences, Physiotherapy and Rehabilitation Department; Eylem Tütün Yümin, PhD, Principal Investigator — BAIBU, Faculty of Health Sciences, Physiotherapy and Rehabilitation Department; Suat Konuk, MD, Principal Investigator — BAIBU, Faculty of Medicine, Department of Chest Diseases
Locations (1):
- Bolu Abant Izzet Baysal University, Faculty of Health Sciences, Physiotherapy and rehabilitation department, Bolu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No